CLINICAL TRIAL: NCT05442307
Title: Boosting General Practice pRescription by Individual Educational Fast Academic Detailing Visits About Asthma
Brief Title: Academic Detailing About Asthma
Acronym: BRIEF-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jón Þór Trærup Andersen, MD, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-2021-709
Record Dates: First submitted 2021-10-06; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Prescription Pattern

STUDY DESIGN:
Intervention Model Description: randomized placebo controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- asthma education (Experimental): The general practices in this arm will receive the education visits about asthma.
  Interventions: Behavioral: asthma education
- Other education (Placebo Comparator): The general practices in this arm will receive an educational visit on another topic (PPI).
  Interventions: Behavioral: Other education

INTERVENTIONS:
Behavioral: asthma education — A 15 minutes (preferable) one-on-one educational visit about asthma treatment. The main points being: Every person with asthma should be treated with inhaled corticosteroids (ICS). Most patients with asthma should be treated with Bufomix Easyhaler either as needed and/or regularly. Patients should not use short-acting bega2-agonist (SABA) unless they use a medium-ICS-dosis.
  Arms: asthma education
Behavioral: Other education — A 15 minutes (preferable) one-on-one educational visit about another topic (NOT asthma).
  Arms: Other education

SUMMARY:
General practices in the Capital Region of Denmark are offered a short educational visit and are randomized to either asthma (intervention) or another topic (control).

The change in prescription pattern from before to after the visit is compared between the intervention and control group.

DETAILED DESCRIPTION:
General practices in the Capital Region of Denmark are offered a short educational visit. They are randomized by address to be offered a visit about either asthma (intervention) or another topic (control).

The prescription pattern of each general practice (as seen by their regional registration number [ydernummer]) who receive a visit is investigated.

The change in prescription pattern from before to after the visit is compared between the intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* General practices in the capital region of denmark, who owns a regional registration number [ydernummer]
* Want a visit
* Have time for a visit within the study period

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change of prescription of inhaled corticosteroids and long-acting beta2-agonist (ICS+LABA) before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of number of adult patients with prescriptions on ICS+LABA between asthma-group and placebo-group.
Difference in change of prescription of ICS and SABA (as monotherapy) before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of number of adult patients with prescriptions on ICS and SABA as monotherapy to adults between asthma-group and placebo-group.

SECONDARY OUTCOMES:
Difference in change of prescription of ICS+LABA before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS+LABA between asthma-group and placebo-group
Difference in change of prescription of ICS+LABA before and after educational visit in one year as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS+LABA between asthma-group and placebo-group as interrupted time series analysis
Difference in change of prescription of ICS+LABA before and after educational visit in one year for each month | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS+LABA between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of prescription of ICS and SABA (as monotherapy) before and after educational visit one year | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS or on SABA as monotherapy to adults between asthma-group and placebo-group.
Difference in change of prescription of ICS and SABA (as monotherapy) before and after educational visit one year as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS or on SABA as monotherapy to adults between asthma-group and placebo-group as interrupted time series analysis
Difference in change of prescription of ICS and SABA (as monotherapy) before and after educational visit one year for each month | one year before and one year after educational visit
  Difference in change of number of adult patients with prescriptions on ICS and on SABA as monotherapy to adults between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of prescription of the Easyhaler Device before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of number of adult patients with prescription on the Easyhaler Device between asthma-group and placebo-group
Difference in change of prescription of the Easyhaler Device before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on the Easyhaler Device between asthma-group and placebo-group
Difference in change of prescription of the Easyhaler Device before and after educational visit as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on the Easyhaler Device between asthma-group and placebo-group as interrupted time series analysis
Difference in change of prescription of the Easyhaler Device before and after educational visit for each month | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on the Easyhaler Device between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of prescription of long-acting muscarinic antagonist (LAMA) before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of number of adult patients with prescription on LAMA between asthma-group and placebo-group
Difference in change of prescription of LAMA before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on LAMA between asthma-group and placebo-group
Difference in change of prescription of LAMA before and after educational visit as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on LAMA between asthma-group and placebo-group
Difference in change of prescription of LAMA before and after educational visit for each month | one year before and one year after educational visit
  Difference in change of number of adult patients with prescription on LAMA between asthma-group and placebo-group analyzed by each month in relation to the visit
Difference in change of cost of each medication group before and after educational visit in a six months period | 6-0 months before and 6-12 months after educational visit
  Difference in change of cost (pharmacy retail price) of SABA, ICS, ICS+LABA, LAMA and ICS+LAMA+LABA to adults between asthma-group and placebo-group
Difference in change of cost of each medication group before and after educational visit in one year | one year before and one year after educational visit
  Difference in change of cost (pharmacy retail price) of SABA, ICS, ICS+LABA, LAMA and ICS+LAMA+LABA to adults between asthma-group and placebo-group
Difference in change of cost of each medication group before and after educational visit as interrupted time series analysis | one year before and one year after educational visit
  Difference in change of cost (pharmacy retail price) of SABA, ICS, ICS+LABA, LAMA and ICS+LAMA+LABA to adults between asthma-group and placebo-group
Difference in change of cost of each medication group before and after educational visit for each month | one year before and one year after educational visit
  Difference in change of cost (pharmacy retail price) of SABA, ICS, ICS+LABA, LAMA and ICS+LAMA+LABA to adults between asthma-group and placebo-group analyzed by each month in relation to the visit

CONTACTS AND LOCATIONS:
Overall Officials: Jon tt Andersen, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- University Hospital Bispebjerg and Frederiksberg, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No